CLINICAL TRIAL: NCT02444325
Title: Group Prenatal Care for Women With Diabetes: A Pilot Randomized Control Trial
Brief Title: Diabetes Group Prenatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Denver Health Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201503174
Record Dates: First submitted 2015-04-27; First posted 2015-05-14 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy; Gestational Diabetes; Type 2 Diabetes
Keywords: group prenatal care; CenteringPregnancy; diabetes
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Prenatal Care (No Intervention): Subjects randomized to routine care will receive their care in the usual diabetic clinic attended by residents and faculty. They will receive consultation with the diabetes educator at diagnosis and as needed. Patients are seen every 2 weeks (or more by provider discretion) until 37 weeks and weekly until delivery. Visits are 10-15 minutes and focus on routine screening tests and review of blood sugar logs/medication titration. Each subject's medical chart will be reviewed for demographics, antenatal management, maternal and neonatal outcomes.
- Group prenatal care (Experimental): Group visits will be held every 2 weeks in a continuous cycle through a four session curriculum. Women will have weekly visits beginning at 37 weeks with traditional prenatal visits on the weeks when the group does not meet. Groups of 4-12 women will meet for two hour visits and much of that time will be spent on pregnancy, behavioral health, diabetes and nutrition education. Groups will be co-facilitated by 2 CenteringPregnancy trained providers at each site and an obstetric provider. Women may be instructed to have additional visits in the traditional clinic at the discretion of the obstetric provider.
  Interventions: Behavioral: Group prenatal care

INTERVENTIONS:
Behavioral: Group prenatal care — Women will receive their prenatal care in a group rather than in the 1:1 traditional manner.
  Arms: Group prenatal care

SUMMARY:
The investigators primary objective is to conduct a pilot randomized trial to determine the effect of group prenatal care on self-care activities in women with diabetes.

DETAILED DESCRIPTION:
Long term, the investigators aim to test the central hypothesis that group prenatal care, compared to traditional prenatal care, will improve glycemic control and, ultimately, maternal and neonatal outcomes in women with type 2 and gestational diabetes. The objective of this proposal is to conduct a pilot randomized trial to determine the effect of group prenatal care on self-care activities, which have been associated with improved glycemic control, in women with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* English (WUMC) or Spanish speaking (DH)
* Type 2 White's Class B diabetes OR gestational diabetes diagnosed by 2-step method < 32 weeks
* Ability to attend group prenatal visit at specified days and times
* Willingness to be randomized
* Randomization at 22 weeks 0 days-32 weeks 0 days
* Ability to give informed consent

Exclusion Criteria:

* Multiple gestation
* Major fetal anomaly
* Serious medical co-morbidity necessitating more care than can be safely provided in group setting, as deemed by medical provider
* Serious psychiatric illness including schizophrenia necessitating more care than can safely be provided in group setting, as deemed by medical provider

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07-06 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
effect of group prenatal care on maternal diabetes self-care activities as measured Diabetes Self-Care Activities Measure | 37-39 weeks gestation
  Determine the effect of group prenatal care on maternal diabetes self-care activities as measured by the Diabetes Self-care Activities Measure and confirmed by percentage of recommended blood glucose values completed on logs since initial study visit.

SECONDARY OUTCOMES:
effect of group prenatal care on perinatal mood as measured by Edinburgh Postnatal Depression Scale | baseline and 4-12 weeks postpartum
  Determine the effect of group prenatal care on perinatal mood as measured by the Edinburgh Postnatal Depression Scale
effect of group prenatal care on perceived social support as assessed by the Social Support Scale | 37-39 weeks
  Determine the effect of group prenatal care on perceived social support through the Social Support Scale
Birthweight | delivery admission
  Determine the effect of group prenatal care on birthweight
Gestational age at delivery | delivery admission
  Determine the effect of group prenatal care on preterm delivery
Mean 3rd trimester fasting blood glucose | baseline through delivery
  Determine the effect of group prenatal care on maternal glycemic control through mean 3rd trimester fasting glucose
Breastfeeding | 4-12 weeks postpartum
  Determine the effect of group prenatal care on initiating breastfeeding
Contraception | 4-12 weeks postpartum
  Determine the effect of group prenatal care on initiating contraception

CONTACTS AND LOCATIONS:
Overall Officials: Methodius G Tuuli, MD, MPH, Study Director — Assistant Professor, Washington University in St. Louis
Locations (2):
- United States (2):
  - Denver Health, Denver, Colorado
  - Washington University in St. Louis, St Louis, Missouri